CLINICAL TRIAL: NCT00538980
Title: A Phase II, Non-Randomized Study of the Use of Desatinib (Sprycel) in Treating Patients With Polycythemia Vera (PV) BMS Protocol Number: CA180-104
Brief Title: Dasatinib in Polycythemia Vera
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to lack of efficacy.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0701008940; CA180-104
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Polycythemia Vera
Keywords: Polycythemia Vera; PV; P Vera
MeSH Terms: conditions — Polycythemia Vera | interventions — Dasatinib

ARMS (1):
- All patients (Experimental): Patients will receive a once-daily oral administration of dasatinib at a dose of 100 mg QD (two 50 mg tablets taken together each day) for the duration of the study with the modifications as indicated. If the platelet count remains above 600,000/microL or the spleen remains enlarged in the absence of leukopenia or other side effects, the dose of dasatinib may be escalated to 120 mg QD (two 50 mg tablets plus one 20 mg tablet taken together each day).
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Patients will receive a once-daily oral administration of dasatinib at a dose of 100 mg QD (two 50 mg tablets taken together each day) for the duration of the study with the modifications as indicated. If the platelet count remains above 600,000/microL or the spleen remains enlarged in the absence of leukopenia or other side effects, the dose of dasatinib may be escalated to 120 mg QD (two 50 mg tablets plus one 20 mg tablet taken together each day).

SUMMARY:
The purpose for conducting this research study is to determine the feasibility of using dasatinib as a treatment for polycythemia vera and to determine the optimum treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be >= 18 years old
2. Performance Status (ECOG) 0-3
3. Previous therapies limited to interferon-alpha, hydroxyurea, anagrelide, and imatinib
4. Patients may have documented resistance or intolerance to interferon-alpha, imatinib, hydroxyurea, or anagrelide, but must have been demonstrated to be phlebotomy dependent requiring 6 or more phlebotomies per year to maintain the target HCT.
5. Patients may have newly diagnosed PV.
6. Patients may have had inadequate phlebotomy control on hydroxyurea or imatinib.
7. Adequate Organ Function

   * Total bilirubin < 2.0 times the institutional Upper Limit of Normal (ULN)
   * Hepatic enzymes (AST, ALT ) ≤ 2.5 times the institutional ULN
   * Serum Na, K+, Mg2+, Phosphate and Ca2+³ Lower Limit of Normal (LLN)
   * Serum Creatinine < 1.5 time the institutional ULN
   * Hemoglobin, Neutrophil count, Platelets, PT, PTT all Grade 0-1
8. Ability to take oral medication: dasatinib tablets may be swallowed whole, or may be ingested as a solution. Dasatinib tablets can be dissolved in juice, and can then be administered through a nasogastric tube.
9. Women of childbearing potential (WOCBP) must have:

   * A negative serum or urine pregnancy test within 72 hours prior to the start of study drug administration
10. Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped.
11. Signed written informed consent including HIPAA according to institutional guidelines

Exclusion Criteria:

1. Patients receiving busulfan within six weeks of Study Day 1.
2. Patients receiving treatment with interferon-alpha within 4 weeks of Study Day 1.
3. Patients receiving treatment with imatinib within 14 days of Study, Day 1.
4. Patients with Grade 3 or 4 cardiac problems as defined by the New York Heart Association Criteria.
5. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable.
6. A malignancy [other than the one treated in this study], which required radiotherapy or systemic treatment within the past 5 years.
7. Concurrent medical condition which may increase the risk of toxicity, including:

   * Pleural or pericardial effusion of any grade
   * Clinically-significant coagulation or platelet function disorder (e.g. known von Willebrand's disease)
8. Cardiac Symptoms, consider the following:

   * Uncontrolled angina, congestive heart failure or MI within (6 months)
   * Diagnosed congenital long QT syndrome
   * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
   * Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
   * Subjects with hypokalemia or hypomagnesemia if it cannot be corrected
9. History of significant bleeding disorder unrelated to cancer, including:

   * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
   * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
   * Ongoing or recent (≤ 3 months) significant gastrointestinal bleeding
10. Concomitant Medications, consider the following prohibitions:

    * Drugs that are generally expected to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib)
    * The concomitant use of H2 blockers or proton pump inhibitors with dasatinib is not recommended. The use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy.
    * Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy
    * Patient agrees that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia.
    * Patient may not be receiving any prohibited CYP3A4 inhibitors
11. Women:

    * Unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or
    * Have a positive pregnancy test at baseline, or
    * Are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04-30 (Actual); Primary Completion 2010-08-25 (Actual); Study Completion 2010-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Slver, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Hematology/Oncology Associates of Rockland, New City, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - The Jones Clinic, Germantown, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 10
Completed | 0
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Effect of Dasatinib on the Platelet Count and the Stabilization of Hematocrit When Restored by Phlebotomy to Normal Range
Description: To evaluate the effect of dasatinib on the platelet count and the stabilization of hematocrit when restored by phlebotomy to normal range (HCT <45% for men, <42% for women). Analysis was not completed because the study was terminated early due to lack of efficacy.
Time Frame: Lab tests will be performed weekly for the first month, then every 2 weeks for months 2 and 3 and monthly thereafter.
Arm/Group | All Patients
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Performance Status and Development of Side Effects and Complications
Description: To determine change in performance status and development of side effects and complications in patients treated under this protocol. Analysis was not completed because the study was terminated early due to lack of efficacy.
Time Frame: Patients will evaluated weekly for the first month, then every two weeks forr months 2 and 3, and monthly thereafter.
Arm/Group | All Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: Changes in Marrow Cellularity, Reticulin and Fibrous Content
Description: To determine changes in marrow cellularity, reticulin and fibrous content. Analysis was not completed because the study was terminated early due to lack of efficacy.
Time Frame: Bone marrow analysis will be performed at baseline and month 6.
Arm/Group | All Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Cytogenetics
Description: To determine change in cytogenetics if initially abnormal. Analysis was not completed because the study was terminated early due to lack of efficacy.
Time Frame: Cytogenetics analysis will be performed at baseline and month 6.
Arm/Group | All Patients
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in JAK2 Allele Burden
Description: To determine if quantitative change in JAK2 expression occurs as measured by quantitative pyrosequencing. Analysis was not completed because the study was terminated early due to lack of efficacy.
Time Frame: JAK2 analysis will be performed at baseline and month 3.
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse events are not included in this report because the data is not available. Every effort was made to retrieve this data from long-term storage, but unfortunately, it could not be obtained.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient went to ER with acute onset of dyspnea with nausea and vomiting. The pt was cyanotic, diaphoretic, and appeared to be in respiratory distress, with elevated WBC. X-Ray showed pulmonary infiltrates. The patient was admitted and later expired.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No